CLINICAL TRIAL: NCT03887988
Title: International, Multicenter, Prospective Registry to Collect Data on Orbital Fractures (OFx), Their Primary and Secondary Treatment and Outcome
Brief Title: Orbital Fractures Registry
Acronym: OFx
Status: Active, not recruiting | Type: Observational
Sponsor: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Other Study IDs: OFx Registry_RP_v.1.0
Record Dates: First submitted 2019-03-18; First posted 2019-03-25 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Orbital Fractures; Blow Out Fracture of Orbit
Keywords: Fracture fixation; Orbital implant; Midface fracture; Diplopia
MeSH Terms: conditions — Orbital Fractures; Diplopia | interventions — Surgical Procedures, Operative; Periodontal Debridement; Conservative Treatment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Orbital Fracture: Patients with dislocated fracture of the inferior and/or medial orbital wall
  Interventions: Procedure: Primary "early" reconstruction; Other: Nonsurgical; Procedure: Primary "delayed" reconstruction; Procedure: Secondary reconstruction

INTERVENTIONS:
Procedure: Primary "early" reconstruction — Primary surgical reconstruction of the fracture within 3 weeks after injury
  Other Names: Operative; Surgical
Other: Nonsurgical — Nonsurgical treatment of fracture
  Other Names: Conservative
Procedure: Primary "delayed" reconstruction — Primary surgical reconstruction of the fracture more than 3 weeks after injury
  Other Names: Operative; Surgical
Procedure: Secondary reconstruction — Second surgical reconstruction of the fracture after a primary reconstruction.
  Other Names: Secondary surgery

SUMMARY:
Approximately 300 patients presenting orbital blow-out fracture will be enrolled prospectively in this registry. All patients, surgically and nonsurgically treated as per standard (routine) of care will be followed-up (FU) within the registry for a period of 6 months.

DETAILED DESCRIPTION:
Approximately 300 patients presenting with a displaced orbital fracture (OFx) in the floor and/or medial wall (blow-out fracture) will be enrolled prospectively in this registry. All patients, surgically and nonsurgical treated will be followed-up (FU) within the registry. FU period for all patients will include assessments post-treatment at 6 weeks, 3 months and 6 months as corresponding with the local standard (routine) visit schedule at each participating clinic.

Data collection includes patient and fracture details, treatment details, functional, clinical and patient-reported outcomes and anticipated or procedure- and implant-related adverse events (ie, complications). Computer Tomography (CT) scans or Cone Beam-CT (CBCT) scans taken as per standard of care will be collected within the registry.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at the time of the injury
* Patients with a dislocated fracture of the inferior and/or medial orbital wall, either

  * Diagnosed at the study site via CT or CBCT within 2 weeks of the date of the injury, OR
  * Who will undergo secondary reconstruction

Exclusion Criteria:

* Bilateral orbital fracture
* Concomitant displaced fracture(s) of the orbital roof or any other area of the orbit
* Concomitant ruptured globe
* Displaced fracture of the malar bone
* Displaced midface fracture
* Displaced nasoorbitoethmoidal (NOE) fracture or complex zygoma fractures
* Presence at the time of enrollment of any disease with influence on eye motility (eg, strabismus, myasthenia gravis, Graves' ophthalmopathy)
* Previous radiotherapy in the orbital region
* Participation in any other medical device or medicinal product study within the previous month(s) that could influence the results of the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years old with displaced fracture of the inferior and/or medial orbital wall (blow-out fractures) that require treatment (either surgically or non-surgically)
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Diplopia | 24 weeks post-treatment
  The degree of diplopia is quantified by measuring the field of single binocular vision, ranging from 0 to 3.
  0: no diplopia
  1. mild (diplopia appears more than 30 degrees from the primary position)
  2. moderate (diplopia appears between 10 and 30 degrees from the primary position)
  3. severe (diplopia appears within 10 degrees from the primary position)

SECONDARY OUTCOMES:
Globe position | 6, 12, 24 weeks post-treatment
  Exo/enophthalmos (in mm) using Naugle or Hertel exophthalmometer Hyper/hypophthalmos: vertical globe displacement is measured as the pupilar height difference (in mm) from the healthy side to the injured side
Visual acuity | 6, 12, 24 weeks post-treatment
  Measured using a visual test chart in healthy and injured sides with and without vision aids.
Extra-ocular mobility | 6, 12, 24 weeks post-treatment
  Follow-my finger test
Patient-reported outcomes | pre-treatment, 6, 12, 24 weeks post-treatment
  AOCMF Injury symptom battery Self-reported diplopia Self-perception of visual acuity, strabismus and symmetry

CONTACTS AND LOCATIONS:
Overall Officials: Eppo B. Wolvius, Prof., Principal Investigator — Department of Oral & Maxillofacial Surgery, Erasmus MC, Rotterdam
Locations (14):
- UC Davis, Sacramento, California, United States
- Germany (2):
  - Medical Center Hamburg Eppendorf, Hamburg
  - Klinikum der LMU München, Munich
- Eramus MC, Rotterdam, Netherlands
- Mayo Hospital, Lahore, Pakistan
- Hamad Medical Corporation, Doha, Qatar
- Emergency Clinical County Hospital of Constanta, Constanța, Romania
- Federal State Budgetary Institution "National Medical and Surgical Center named after N.I. Pirogov" of the Ministry of Healthcare of the Russian Federation, Moscow, Russia
- Clinic for Maxillofacial Surgery, University of Belgrade, Belgrade, Serbia
- King Edward VIII Hospital, Durban, South Africa
- Spain (2):
  - Hospital Vall d' Hebron, Barcelona, Catalonia
  - 12 de Octubre University Hospital, Madrid, Madrid
- Uppsala University Hospital, Uppsala, Sweden
- Universitaetsspital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Strabbing EM; OFx Registry Study Group; Wolvius EB. Surgical versus non-surgical management of orbital fractures: study protocol for evidence generation of a prospective multicentre observational cohort registry. BMJ Open. 2025 Jul 30;15(7):e100508. doi: 10.1136/bmjopen-2025-100508. PMID 40738644